CLINICAL TRIAL: NCT02886143
Title: Effect of Active vs. Passive Voiding Trials on Time to Patient Discharge, Rate of Urinary Tract Infection, and Rate of Urinary Retention: a Randomized, Controlled Clinical Trial
Brief Title: Effect of Active vs. Passive Voiding Trials on Time to Discharge, Urinary Tract Infection, and Urinary Retention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Tracey Krupski, MD, Vice Chair, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18345
Record Dates: First submitted 2016-07-31; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Urinary Retention; Urinary Tract Infections
MeSH Terms: conditions — Urinary Retention; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Voiding Trial (instillation of sterile saline) (Experimental): Patients randomized to receive an active voiding trial will have the bladder filled with 250-400 cc of sterile saline (or until the bladder was full) via the lumen of the urinary catheter before the urinary catheter is removed. The patient will then be immediately assisted to void. Physician teams will follow a standardized algorithm for the management of urinary retention arising during the study.
  Interventions: Procedure: Active Voiding Trial
- Passive Voiding Trial (Active Comparator): For patients randomized to receive a passive voiding trial, the urinary catheter will be removed, the bladder will fill with urine naturally, and the patient will be assisted to void when he or she reports the urge. To ensure uniformity in the intervention, all voiding trials in the study will be supervised by an experienced nurse who will ensure that the protocol is followed.
  Interventions: Procedure: Passive Voiding Trial

INTERVENTIONS:
Procedure: Active Voiding Trial — Nursing protocol:
  1. Instill 250-400 cc of STERILE SALINE via the lumen of the Foley catheter into the bladder via gravity drainage or slow push
  2. Clamp the Foley
  3. Deflate the catheter balloon and remove the catheter from the bladder.
  4. Record the amount of saline that was instilled into the bladder.
  5. Immediately assist the patient to void. Report the amount instilled and the amount voided to the physician within one hour a. Unless the patient reports extreme bladder fullness or pain, give the patient one hour to urinate
  7. If the patient fails the voiding trial, the physician will decide to do in and out catheterization or place a new Foley catheter
  Arms: Active Voiding Trial (instillation of sterile saline)
Procedure: Passive Voiding Trial — Nursing protocol:
  1. Deflate the catheter balloon and remove the catheter from the bladder.
  2. Record the time that the catheter was removed and the time the patient is due to void (approximately 6 hours).
  3. 5. If the patient has not voided within 5 hours, assist the patient to try to void.
  6. If the patient is unable to void, is only voiding in small amounts, or reports fullness or abdominal pain, perform a bladder scan.
  7. If the patient has not voided after 6 hours, report this to the physician along with the results of the bladder scan 8. The physician will decide to do in and out catheterization or place a new Foley catheter
  Arms: Passive Voiding Trial

SUMMARY:
Urinary retention is a common problem, particularly in hospitalized patients. When a Foley catheter is removed, a patient must be monitored for urinary retention. The usual method is a passive voiding trial where the catheter is removed, the bladder fills with urine and the patient is monitored for voiding over approximately 6 hours. Another option is an active voiding trial where the bladder is filled with saline before the catheter is removed and the patient is immediately assisted to void. This study seeks to determine the effect of active vs passive voiding trials on time to hospital discharge, rate of urinary tract infections, and rate or urinary retention in the general hospitalized population.

DETAILED DESCRIPTION:
The intervention to be tested is an active voiding trial, where the bladder is filled with saline before the catheter is removed and the patient is immediately assisted to void.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of three hospital units at the University of Virginia (5 Central, 6 West, or the Short Stay Unit)
* Patient has a Foley urethral catheter in place
* The physician has ordered the Foley urethral catheter to be discontinued
* 18 years of age and older

Exclusion Criteria:

* Age less than 18 years
* Prisoners
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
time from removal of Foley catheter until hospital discharge | approximately one day
  time from removal of the Foley catheter until the patient physically leaves the hospital

SECONDARY OUTCOMES:
urinary tract infection | within 2 weeks of hospital discharge
  urinary tract infection within 2 weeks of hospital discharge based on the National Surgical Quality Improvement Program (NSQIP) definition (one of two of the following):
  1. One of the following: (fever (>38 C), urgency, frequency, dysuria, or suprapubic tenderness) AND urine culture of >10^5 colonies/mL urine with no more than 2 species of organisms
  2. Two of the following (fever (>38 C), urgency, frequency, dysuria, or suprapubic tenderness) AND any of the following: (dipstick test positive for leukocyte esterase and/or nitrite, pyuria (>10 white blood cells (WBC)/mL or >3 WBC/hpf of unspun urine), organisms seen on Gram stain of unspun urine, two urine cultures with repeated isolation of the same uropathogen with >10^2 colonies/mL urine in non-voided specimens, urine culture with <10^5 colonies/mL urine of single uropathogen in patient being treated with appropriate antimicrobial therapy, physician's diagnosis, physician institutes appropriate antimicrobial therapy)
Urinary retention | within 2 weeks of hospital discharge
  inability to urinate requiring urethral catheterization within 2 weeks of hospital discharge. This will be determined by asking the patient the number of times he or she has had a urethral catheter inserted in the 2 weeks since the catheter was removed

CONTACTS AND LOCATIONS:
Overall Officials: Tracey L Krupski, MD, MPH, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mills JT, Rapp DE, Shaw NM, Hougen HY, Agard HE, Case RM Jr, McMurry TL, Schenkman NS, Krupski TL. Effect of active versus passive void trials on time to patient discharge, urinary tract infection, and urinary retention: a randomized clinical trial. World J Urol. 2020 Sep;38(9):2247-2252. doi: 10.1007/s00345-019-03005-0. Epub 2019 Nov 15. PMID 31732771